CLINICAL TRIAL: NCT03258255
Title: Comparison of Analgesic Efficiency of Pudendal Nerve Block and Penil Block for Circumsion in Children
Brief Title: Analgesic Efficiency of Pudendal Nerve Block Versus Penil Block for Circumsion in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ayse Cigdem Tutuncu, assoc prof, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 242893
Record Dates: First submitted 2017-08-20; First posted 2017-08-23 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Postoperative Analgesia
MeSH Terms: interventions — Circumcision, Male

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pudendal block group in circumcision (Active Comparator): Nerve stimulated pudendal nerve block performed under general anesthesia
  Interventions: Procedure: penil or pudendal nerve block in circumcision
- Penil block group in circumcision (Active Comparator): Penil block performed by surgeon under general anesthesia
  Interventions: Procedure: penil or pudendal nerve block in circumcision

INTERVENTIONS:
Procedure: penil or pudendal nerve block in circumcision — regional analgesia methods during the circumsion nerve stimulator guided pudendal block performed by anesthesiologist/ penil block performed by surgeon before circumcision

SUMMARY:
The aim of this prospective randomized study is to assess the analgesic efficacy of Pudendal block compared with penil block for pediatric patients undergoing circumsion concerning postoperative analgesic consumption within 24 hours.

DETAILED DESCRIPTION:
In this prospective study, patients will be randomized into 2 groups, either receiving penil Block( PNL) or nerve stimulator-guided Pudendal Nerve Block(PNB). Analgesic consumption will be assessed during the first 24 hours postoperatively. The "CHEOPS pain scale" will use to assess postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

ASA I-II patients, aged 1-12 years old patient undergoing circumcision,

Exclusion Criteria:

history of local anesthetics's allergy, infection at the injection side, anatomical abnormalities, coagulopaty, bleeding disease, liver disease

Ages: 1 Year to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Postoperative pain evaluatiom | 24 hour
  CHEOPS pain scale

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cyna AM, Middleton P. Caudal epidural block versus other methods of postoperative pain relief for circumcision in boys. Cochrane Database Syst Rev. 2008 Oct 8;2008(4):CD003005. doi: 10.1002/14651858.CD003005.pub2. PMID 18843636